CLINICAL TRIAL: NCT00245167
Title: TLR's, Nitric Oxide and Chronic Lung Disease: Any Connections?
Brief Title: Possible Relation of Toll-Like Receptors and Nitric Oxide to Chronic Lung Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1316; R01HL070560 (NIH)
Record Dates: First submitted 2005-10-26; First posted 2005-10-27 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-03

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases

INTERVENTIONS:
Procedure: Tracheal Aspirate Fluid

SUMMARY:
The first objective of this study is to determine if increased expression of one or more members of the toll-like receptor (TLR) family of receptors that are found on inflammatory cells (present in the airway) precede development of chronic lung disease (CLD) of prematurity. The study will also determine if there is a significant correlation between TLRs and the severity of CLD. The second objective of this study is to determine the impact of c-administration of inhaled nitric oxide (INO) on TLR expression in infants at risk of developing CLD or with early CLD.

DETAILED DESCRIPTION:
BACKGROUND:

This study will examine the role of two members in the family of transmembrane receptors, TLRs, found on leukocytes and other cells that are upregulated in response to endotoxin and other stimuli. These substances transfer the signals that propagate inflammation and production of inflammatory cytokines. CLD of prematurity is characterized by early (first week of life) evidence of lung airway inflammation. It is unknown if TLR family members propagate this pathway.

DESIGN NARRATIVE:

This study will involve saving weekly tracheal aspirate fluid samples obtained with routine airway toilet in infants less than or equal to 1250 gm birth weight, who are admitted to a Neonatal Intensive Care unit requiring assisted ventilation via an endotracheal tube. The waste sample will be collected with the cellular contents separated by centrifugation and placed on Trizol reagent after obtaining a cell count. Later extraction and batch analysis of TLR, mRNA, and proteins as well as mRNA and protein for housekeeping genes will be performed. Immunohistochemistry will also be used to semi-quantitate the samples. Samples will be obtained in the first one to two days, and again at the end of the first week of life. In infants who were also participating in the related "Low Dose INO in CLD of Prematurity" study, in which tracheal aspirate samples were collected, when the code is broken to determine who received nitric oxide versus placebo, the second aim of the study will be carried out: to determine the impact, if any, of INO.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight less than 1250 gm
* Requiring assisted ventilation

Exclusion Criteria:

* Moribund condition
* Major pulmonary or cardiovascular associated anomaly

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120
Dates: Start 2002-01; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William E. Troug, MD, Principal Investigator — Children's Mercy Hospital & Clinic
Locations (2):
- United States (2):
  - Children's Mercy Hospital & Clinic, Kansas City, Missouri
  - Children's Hospital and Regional Medical Center (Seattle), Seattle, Washington